CLINICAL TRIAL: NCT02327923
Title: Intraoperative Lidocaine Infusion vs. Esmolol Infusion for Postoperative Analgesia in Laparoscopic Cholecystectomy: a Randomized Clinical Trial
Brief Title: Intraoperative Lidocaine Infusion vs. Esmolol Infusion for Postoperative Analgesia in Laparoscopic Cholecystectomy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: B.P. Koirala Institute of Health Sciences (Other)
Responsible Party: Principal Investigator, Joshan Lal Bajracharya, Junior resident, B.P. Koirala Institute of Health Sciences
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: IERB/284/014
Record Dates: First submitted 2014-10-12; First posted 2014-12-31 (Estimated); Last update posted 2018-11-30 (Actual); Status verified 2018-11

CONDITIONS: Gall Stone Disease
Keywords: Laparoscopic cholecystectomy; lidocaine infusion; Esmolol infusion; Postoperative opioid consumption; Multimodal analgesia
MeSH Terms: interventions — Lidocaine; esmolol; Acetaminophen; Propofol; Fentanyl; Vecuronium Bromide; Atropine; Ephedrine; Morphine; Ketorolac; Ondansetron; Bupivacaine; Tramadol; Neostigmine; Glycopyrrolate

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lidocaine (Active Comparator): Intravenous bolus administration of lidocaine at the time of induction followed by infusion till the last suture.
  Interventions: Drug: Lidocaine; Drug: Paracetamol; Drug: Propofol; Drug: Fentanyl; Drug: Vecuronium; Drug: Atropine; Drug: Ephedrine; Drug: Morphine; Drug: Ketorolac; Drug: Ondansetron; Drug: Bupivacaine; Drug: Tramadol; Drug: Neostigmine; Drug: Glycopyrrolate
- Esmolol (Active Comparator): Intravenous bolus administration of esmolol at the time of induction followed by infusion till the last suture.
  Interventions: Drug: Esmolol; Drug: Paracetamol; Drug: Lidocaine; Drug: Propofol; Drug: Fentanyl; Drug: Vecuronium; Drug: Atropine; Drug: Ephedrine; Drug: Morphine; Drug: Ketorolac; Drug: Ondansetron; Drug: Bupivacaine; Drug: Tramadol; Drug: Neostigmine; Drug: Glycopyrrolate

INTERVENTIONS:
Drug: Lidocaine — Lidocaine intravenous 1.5mg/kg IV bolus at the time of induction followed by IV infusion @ 1.5 mg/kg/hr till the last suture.
  Other Names: Lignocaine, Xylocaine
  Arms: Lidocaine
Drug: Esmolol — Esmolol intravenous bolus 0.5 mg/kg at the time of induction followed by infusion @ 5-15 microgram/kg/min till the last suture.
  Arms: Esmolol
Drug: Paracetamol — Inj. Paracetamol 1 gm IV at the time of induction
Drug: Lidocaine — Inj. Xylocaine 2% 3 ml will be infiltrated in skin in all port sites prior to incision.
  Other Names: Xylocaine
Drug: Propofol — Inj. Propofol 2- 2.5 mg/kg will be given for induction
Drug: Fentanyl — Inj fentanyl 1.5mg/kg will be given at the time of induction.
Drug: Vecuronium — Inj Vecuronium 0.1mg/kg will be given at induction and for maintenance.
Drug: Atropine — Inj Atropine 0.4 mg IV will be given for bradycardia (HR < 50/min)
Drug: Ephedrine
Drug: Morphine
Drug: Ketorolac
Drug: Ondansetron
Drug: Bupivacaine — Inj. Bupivacaine 0.25% 10 ml will be infiltrated at incision site after closure.
Drug: Tramadol — Inj tramadol 50 mg IV will be given on SOS basis in ward.
Drug: Neostigmine — 50 mcg/kg for reversal of residual neuromuscular blockade
Drug: Glycopyrrolate — 10 mcg/kg with neostigmine

SUMMARY:
Comparison of intraoperative infusion of lidocaine and esmolol in the postoperative requirement of opioid for postoperative pain management after laparoscopic cholecystectomy to decrease opioid related side effects and enhance postoperative recovery with multimodal analgesia approach.

DETAILED DESCRIPTION:
Postoperative pain after abdominal surgery includes many forms of distress, such as spontaneous pain at rest; pain during movement, including that of respiration; and visceral pain arising from damage to internal organs during surgery. Acute pain after laparoscopic cholecystectomy is complex in nature. The pain pattern does not resemble pain after other laparoscopic procedures, suggesting that analgesic treatment might be procedure specific and multimodal. Three components have been described: incisional pain as dominant, visceral deep pain, and shoulder referred pain. Opioids are most commonly used for postoperative analgesia in laparoscopic cholecystectomy. However, they can be associated with many side effects and delayed discharge. In addition, opioids do not offer the quality of postoperative pain relief that one would expect, probably because of the pain specific to laparoscopic cholecystectomy. A single agent is unlikely to treat all three types of pain. Therefore a multimodal approach will be required.

Low-dose IV lidocaine is easy to administer, has well-established analgesic, anti-hyperalgesic, and anti-inflammatory effects, and has minimal toxicity in commonly studied doses (typically 1.5-3 mg/kg/h). Because postoperative pain is to a large extent an inflammatory phenomenon, administration of systemic local anesthetics, which have inflammatory modulatory properties, could significantly reduce pain and therefore allow more rapid discharge. Lidocaine has an excellent safety record when administered by low-dose infusion. In addition, intravenous lidocaine is an effective modality for treating visceral pain.

Esmolol has been proposed as an alternative to intraoperative use of opioids, and found to facilitate the fast-tracking process and speed home-readiness of patients undergoing outpatient surgery. The various mechanisms of opioids dose sparing with concomitant use of β-adrenergic antagonist have been proposed from time to time such as suppression of stress hormones and pro-inflammatory cytokines, alteration of hepatic drug metabolism, activation of G-coupled proteins in cell membrane, central analgesia and so on but nothing conclusive has been established as yet.

After pre operative evaluation, patients will be premedicated with oral diazepam (0.1-0.2 mg/kg) at the night before and 2 hours before surgery. Informed consent will be obtained from all patients. Patients will be instructed during pre-anaesthetic visit about the use of the visual analogue scale (0-10 cm) where 0 is no pain and 10 is worst imaginable excruciating pain. They will also be informed that they will be asked their pain (VAS score) with its character during first 24 hrs after the surgery.

Both the patient and the investigator observing the outcome will be blinded about assignment of patient group during the study. The investigator will not enter the operating room but will be responsible for data collection in post operative period and data analysis. On arrival of patients in the preoperative holding area, they will be randomly assigned into any of two groups using computer generated random number. Details of group assignment and case number will be kept in a set of sealed opaque envelope. The anesthesia staff will open the envelope and prepare drugs accordingly. The attending anesthesiologist will not be involved in the data collection and analysis, and will follow the standard general anaesthesia protocol during the study.

On arrival to operating room, standard monitoring will be established and baseline heart rate, non-invasive B.P, oxygen saturation and bispectral index (BIS) value (Covidien) will be recorded. A peripheral vein will be cannulated for administration of IV fluid with 18 G cannula Patient will be preoxygenated using 100% oxygen for 3 minutes.

General anesthesia will be induced with IV fentanyl 1.5 µg/kg , propofol 2-2.5 mg/kg till cessation of verbal response and tracheal intubation facilitated with vecuronium 0.1mg/kg IV. The lungs will be mechanically ventilated with a 50% mixture of air in oxygen to maintain ETCO2 between 35 to 45 mm of Hg. At induction, lidocaine group (L group) patients will receive 1.5 mg/kg of lidocaine IV bolus. The lidocaine infusion (B-Braun) of 1.5 mg/kg/h will be started immediately after induction of anesthesia. The esmolol group (E group) will receive an IV bolus 0.5 mg/kg at induction followed by continuous infusion (B-Braun) of esmolol (5-15 μg/kg/min) and titrated to maintain the heart rate within 25% of the baseline value. Inj. paracetamol 1 gm IV infusion will be started after induction and given over 15 min.

Anesthesia will be maintained in all groups with isoflurane adjusted upto 2.5% to maintain MAP within 20% of baseline and BIS value between 50 to 60. An orogastric tube will be inserted in every patient before surgical incision. No supplemental opioids will be used during surgery. Supplemental neuromuscular blockade will be achieved with vecuronium IV bolus doses after observing curare notch in capnometry. Inj. ketorolac 30 mg IV and ondansetron 4mg (0.1mg/kg) IV will be given after removal of gall bladder. Any episode of intraoperative hypotension (MAP lower than 65 mm Hg) and bradycardia (heart rate < 50 bpm) will be treated with ephedrine 5 mg and atropine 0.4 mg IV respectively.

Patient position and monitoring

Hasson surgical technique will be used. Each port site will be infiltrated with 3ml of 2% lidocaine before incision. Pneumoperitoneum will be achieved with carbon dioxide. Patients will be positioned in 30 degrees reverse trendelenburg position and tilted toward the left slowly. Non-invasive blood pressure assessment, oximetry, ECG and end tidal CO2 will be continually monitored during the anesthesia. During pneumoperitoneum, controlled ventilation will be adjusted to maintain ETC02 between 35 to 45 mm of Hg. Intra-abdominal pressure will be kept below 15 mm of Hg during laparoscopy.

At the end of surgery, patients will be returned to a supine position and the carbon dioxide left in the peritoneal cavity will be expelled by slow abdominal decompression. Isoflurane will be discontinued after the last skin suture, and the lignocaine or esmolol infusions will also be stopped at completion of surgery. 10 ml of 0.25% Bupivacaine will be infiltrated in the incision site.

Residual neuromuscular block will be reversed with neostigmine 0.05 mg/kg IV and glycopyrrolate 0.01 mg/kg IV. Thorough gastric and oropharyngeal suctioning will be done. Then, orogastric tube will be removed before endotracheal extubation. Trachea will be extubated on the operating table. Then, the patient will be transferred to the postanesthesia care unit.

Postoperative Care and observation In PACU, non-invasive blood pressure, heart rate, respiration, and temperature will be monitored by nurses unaware of the study. Pain at awakening will be noted using VAS scale. Pain including its character will be assessed at rest and on movement by a VAS every 30 min by the investigator and by nurses on SOS basis on patient's request. If the VAS for pain is more than 3 at rest, morphine 1 mg IV and Tramadol 50 mg IV will be administered in PACU and in ward respectively and repeated on SOS basis. It will be stopped if any adverse effects noticed which will include increased sleepiness, respiratory depression (SPO2 < 90%, R.R < 8 per minute). Metoclopramide 10 mg IV will be administered for grade 3 & 4 PONV.

In the investigators institution, no step-down high dependency unit is available and patients will be transferred to ward directly from the PACU and following outcome parameters will be observed at 2, 6, 8, 12 and 24 h after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Adult female patients of ASA physical status I or II, between age of 18 to 60 years undergoing elective laparoscopic cholecystectomy under general anaesthesia.

Exclusion Criteria:

* Refusal to give consent.
* ASA physical status III or more.
* Inability to comprehend pain assessment score or severe mental impairment.
* Difficult intubation.
* Pregnancy.
* Morbid obesity.
* History of epilepsy.
* History of allergy to any drug used in the study.
* History of ongoing use of opioids or beta adrenergic receptor antagonists.
* Baseline heart rate less than 50 beats per minute.
* Presence of pain immediately before surgery.
* Chronic pain other than gall stone disease.
* Gastrointestinal ulceration, bleeding disorder.
* Peritonitis (including previous), perforated gall bladder, severe acute cholecystitis, known to have choledocholithiasis.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2016-02 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Opioid (morphine equivalent) requirement in the first 24 h postoperatively | up to 24 hours postoperatively
  total morphine consumed in the first 24 h postoperatively

SECONDARY OUTCOMES:
Visual analogue scale (VAS) scores for pain severity | up to 24 hours postoperatively
  Pain at rest and with cough or movement using the VAS scale during first 24 h (at PACU and ward). VAS scale consist of a line with 10 cm length, where "0" is no pain and "10" is worst pain patient can imagine.
Incidence of postoperative nausea and vomiting (PONV). | up to 24 hours postoperatively
  Incidence of postoperative nausea and vomiting (PONV) in the first 24 h using PONV scoring.
Time to first voiding | up to first 24 hours postoperatively
Sedation score using Ramsay Scale. | up to 24 hours postoperatively
  Sedation score using Ramsay Scale during first 24 h postoperatively.
Patient satisfaction following Laparoscopic cholecystectomy | at 24 hours postoperatively
  Patient satisfaction following LC using Likert Satisfaction Scale at 24 h following surgery
Time to first perception of pain | up to 24 hours postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Asish Subedi, MD, Study Director — B.P. Koirala Institute of Health Sciences
Locations (1):
- BP Koirala Institute of Health Sciences, Dharān, Sunsari District, Nepal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Collard V, Mistraletti G, Taqi A, Asenjo JF, Feldman LS, Fried GM, Carli F. Intraoperative esmolol infusion in the absence of opioids spares postoperative fentanyl in patients undergoing ambulatory laparoscopic cholecystectomy. Anesth Analg. 2007 Nov;105(5):1255-62, table of contents. doi: 10.1213/01.ane.0000282822.07437.02. PMID 17959952
- [Background] Lauwick S, Kim DJ, Michelagnoli G, Mistraletti G, Feldman L, Fried G, Carli F. Intraoperative infusion of lidocaine reduces postoperative fentanyl requirements in patients undergoing laparoscopic cholecystectomy. Can J Anaesth. 2008 Nov;55(11):754-60. doi: 10.1007/BF03016348. PMID 19138915
- [Background] McCarthy GC, Megalla SA, Habib AS. Impact of intravenous lidocaine infusion on postoperative analgesia and recovery from surgery: a systematic review of randomized controlled trials. Drugs. 2010 Jun 18;70(9):1149-63. doi: 10.2165/10898560-000000000-00000. PMID 20518581
- [Background] Marret E, Rolin M, Beaussier M, Bonnet F. Meta-analysis of intravenous lidocaine and postoperative recovery after abdominal surgery. Br J Surg. 2008 Nov;95(11):1331-8. doi: 10.1002/bjs.6375. PMID 18844267
- [Background] Lee MH, Chung MH, Han CS, Lee JH, Choi YR, Choi EM, Lim HK, Cha YD. Comparison of effects of intraoperative esmolol and ketamine infusion on acute postoperative pain after remifentanil-based anesthesia in patients undergoing laparoscopic cholecystectomy. Korean J Anesthesiol. 2014 Mar;66(3):222-9. doi: 10.4097/kjae.2014.66.3.222. Epub 2014 Mar 28. PMID 24729845
- [Background] Lopez-Alvarez S, Mayo-Moldes M, Zaballos M, Iglesias BG, Blanco-Davila R. Esmolol versus ketamine-remifentanil combination for early postoperative analgesia after laparoscopic cholecystectomy: a randomized controlled trial. Can J Anaesth. 2012 May;59(5):442-8. doi: 10.1007/s12630-012-9684-x. Epub 2012 Mar 2. PMID 22383085
- [Background] Ozturk T, Kaya H, Aran G, Aksun M, Savaci S. Postoperative beneficial effects of esmolol in treated hypertensive patients undergoing laparoscopic cholecystectomy. Br J Anaesth. 2008 Feb;100(2):211-4. doi: 10.1093/bja/aem333. Epub 2007 Nov 23. PMID 18037672
- [Derived] Bajracharya JL, Subedi A, Pokharel K, Bhattarai B. The effect of intraoperative lidocaine versus esmolol infusion on postoperative analgesia in laparoscopic cholecystectomy: a randomized clinical trial. BMC Anesthesiol. 2019 Nov 4;19(1):198. doi: 10.1186/s12871-019-0874-8. PMID 31684867